CLINICAL TRIAL: NCT01959035
Title: Interventional, Open-label, Flexible-dose Extension Study of Aripiprazole Once-monthly in Patients With Schizophrenia
Brief Title: Aripiprazole Once-monthly in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14724B; 2012-003239-47 (EudraCT Number)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole once-monthly (Experimental)
  Interventions: Drug: Aripiprazole once-monthly

INTERVENTIONS:
Drug: Aripiprazole once-monthly — 400 or 300 mg/month; 6 intramuscular (IM) injections starting at baseline
  Other Names: Abilify Maintena®

SUMMARY:
To obtain information on the safety, tolerability and effectiveness of aripiprazole once-monthly in a manner consistent with its intended use in everyday clinical practice in patients with schizophrenia who completed Study 14724A / NCT01795547.

ELIGIBILITY:
Patients will be recruited among those who complete treatment with aripiprazole in Study 14724A / NCT01795547.

Inclusion Criteria:

* The patient is judged to potentially benefit from 24-week treatment with aripiprazole once-monthly according to the clinical opinion of the investigator.
* The patient agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

* The patient has been diagnosed with a primary psychiatric disorder other than schizophrenia during Study 14724A / NCT01795547.
* The patient has a clinically significant unstable illness diagnosed during Study 14724A / NCT01795547.
* The patient is at significant risk of harming himself/herself or others according to the investigator's judgement or according to Columbia-Suicide Severity Rating Scale (C-SSRS).
* The patient has a disease or takes medication that could, in the investigator's opinion, interfere with the assessments of safety, tolerability or efficacy, or interfere with the conduct or interpretation of the study.
* The patient has one or more clinical laboratory test values outside the reference range, based on the blood or urine samples taken during the conduct of Study 14724A / NCT01795547 that are, in the investigator's opinion, of potential risk to the patient's safety.
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- US006, San Diego, California, United States

REFERENCES:
- See also: EMA EudraCT Results: 2012-003239-47 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-003239-47/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole Once-monthly: Aripiprazole once-monthly: 400 or 300 mg/month depending on the last dose that they had received in Study 14724A; 6 intramuscular (IM) injections starting at baseline
Period: Overall Study
Arm/Group | Aripiprazole Once-monthly
Started | 88
Completed | 77
Not Completed | 11
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Other (no primary reason given) | 1

BASELINE CHARACTERISTICS:
Population: Demographic data is based on all patients who received at least one dose of IMP in Study 14724B.
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of treatment emergent adverse events (TEAEs).
Time Frame: Up to 24 weeks and 4-week safety follow up
Population: Safety data is based on all patients who received at least one dose of investigational medicinal product (IMP) in Study 14724B.
Measure: Number; unit: number of events
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 88
number of events | 65

2. Secondary Outcome: Change From Baseline to Week 24 in SWN-S Total Score
Description: The Subjective Well-Being under Neuroleptic Treatment - Short Version (SWN-S) is a patient-rated scale designed to measure subjective effects of neuroleptic drugs to psychopathology, quality of life, and compliance over the past 7 days. The 20 items (10 positive and 10 negative statements) are grouped in 5 subscales (mental functioning, self-control, physical functioning, emotional regulation and social integration). Each subscale contains 4 items. Each item was rated on a six-point Likert scale, from not at all to very much. A score was calculated for each subscale, and the total score ranged from 20 to 120, where the higher score indicated better well-being.
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for SWN-S total score was based on the 75 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 75
units on a scale | 0.19 [-2.08 to 2.45]

3. Secondary Outcome: Change From Baseline to Week 24 in CGI-S Score
Description: Clinical Global Impression - Severity of Illness (CGI-S) score provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (normal - not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for CGI-S score was based on the 78 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 78
units on a scale | -0.10 [-0.26 to 0.06]

4. Secondary Outcome: Change From Baseline to Week 24 in QLS Total Score
Description: The Quality of Life Scale (QLS) is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). Definitions were provided for 4 anchor points of the 7 points. Each item had a brief description of the judgement to be made and a set of suggested probes for the clinician. The total score was calculated as the sum of all 21 items giving a range of 0 to 126, where the higher score indicated normal or unimpaired functioning.
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for QLS total score was based on the 78 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 78
units on a scale | 2.32 [-1.21 to 5.85]

5. Secondary Outcome: Change From Baseline to Week 24 in the 'Common Objects and Activities' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Common Objects and Activities domain score was calculated as the sum of 2 items (numbers 18 and 19) giving a range of 0 to 12, where the higher score indicated less unimpaired functioning
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for 'Common Objects and Activities' QLS domain score was based 78 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 78
units on a scale | 0.21 (1.29)

6. Secondary Outcome: Change From Baseline to Week 24 in the 'Intrapsychic Foundations' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Intrapsychic Foundations domain score was calculated as the sum of 7 items (numbers 13 to 17 and 20 and 21) giving a range of 0 to 42, where the higher score indicated less unimpaired functioning
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for 'Intrapsychic Foundations' QLS domain score was based on the 78 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 78
units on a scale | 0.72 (5.03)

7. Secondary Outcome: Change From Baseline to Week 24 in the 'Interpersonal Relations' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Interpersonal Relations domain score was calculated as the sum of 8 items (numbers 1 to 8) giving a range of 0 to 48, where the higher score indicated less unimpaired functioning.
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for 'Interpersonal Relations' QLS domain score was based on the 78 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 78
units on a scale | 0.58 (6.54)

8. Secondary Outcome: Change From Baseline to Week 24 in the 'Instrumental Role' QLS Domain Score
Description: The QLS is a clinician-rated scale designed to assess deficit symptoms of schizophrenia and functioning during the preceding 4 weeks. The QLS consists of 21 items in 4 domains: Interpersonal Relations (eight items), Instrumental Role (four items), Intrapsychic Foundations (seven items), and Common Objects and Activities (two items). Each item was rated on a 7-point scale, from 0 (severe impairment) to 6 (normal or unimpaired functioning). The Instrumental Role domain score was calculated as the sum of 4 items (numbers 9 to 12) giving a range of 0 to 24, where the higher score indicated less unimpaired functioning.
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for 'Instrumental Role' QLS domain score was based on the 78 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 78
units on a scale | 0.42 (4.54)

9. Secondary Outcome: Change From Baseline to Week 24 in the TooL Total Score
Description: Tolerability and Quality of Life (TooL) is a patient-rated scale developed to measure the impact of side-effects on the quality of life in patients treated with antipsychotic medication. The TooL consists of 8 domains: mood (worry-upset), function capabilities, fatigue-weakness, weight gain, stiffness-tremor, physical restlessness, sexual dysfunction, and dizziness-nausea. Each domain was rated on a four-point scale from 1 (no impact) to 4 (maximum impact). Total scores ranged from 8 (no impact) to 32 (maximum impact).
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for TooL total score was based on the 75 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 75
units on a scale | -0.47 [-1.16 to 0.22]

10. Secondary Outcome: Change From Baseline to Week 24 in the WoRQ Total Score
Description: The Readiness for Work Questionnaire (WoRQ) is a clinician-rated scale designed to measure a schizophrenic patient's ability to work. The WoRQ consists of 8 items: the clinician had to rate 7 statements and answer 1 question. The statements were rated on a four-point scale, from 'strongly agree', 'agree', 'disagree' or 'strongly disagree' based on all material available (for example, personal notes, medical records, input from other health professionals, family members or caregivers); and in the final item, the clinician had to indicate if the patient was ready for work or not (by indicating either 'yes' or 'no'). Possible total scores range from 4 to 28. Lower WoRQ total scores indicate better functioning.
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for WoRQ total score was based on the 77 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 77
units on a scale | -0.53 [-1.21 to 0.15]

11. Secondary Outcome: Change From Baseline to Week 24 in ASEX Total Score
Description: The Arizona Sexual Experience Scale (ASEX) is a five-item, patient-rated scale that evaluates a patient's recent sexual experiences. The ASEX is used to identify individuals with sexual dysfunction. Patients were asked to assess their own experiences over the last week (for example, "How strong is your sex drive?", "Are your orgasms satisfying?") and respond on a six-point scale for each item. Possible total scores range from 5 to 30. Higher ASEX total scores indicate more sexual dysfunction (hypofunction).
Time Frame: Baseline and Week 24
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 24, the analysis for ASEX total score was based on the 75 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 75
units on a scale | -0.42 [-1.74 to 0.91]

12. Secondary Outcome: Patients Categorised As Sexually Dysfunctional Measured at Week 24 on the ASEX Scale
Description: The Arizona Sexual Experience Scale (ASEX) is a five-item, patient-rated scale that evaluates a patient's recent sexual experiences. The ASEX is used to identify individuals with sexual dysfunction. Patients were asked to assess their own experiences over the last week (for example, "How strong is your sex drive?", "Are your orgasms satisfying?") and respond on a six-point scale for each item. Possible total scores range from 5 to 30. Higher ASEX total scores indicate more sexual dysfunction (hypofunction). The presence of sexual dysfunction based on the ASEX scale was defined as an ASEX total score of ≥19, or a score of ≥5 on any item, or a score of ≥4 on any 3 items.
Time Frame: Week 24
Population: This analysis is based on all patients who received at least one dose of IMP in Study 14724B (APTS). At Week 24, the analysis for the number of patients categorised as sexually dysfunctional was based on the 75 patients who had a measure for this outcome
Measure: Number; unit: participants
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 75
participants | 31

13. Secondary Outcome: Change From Baseline to Week 12 in SWN-S Total Score
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for SWN-S total score was based on the 82 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | -1.57 [-4.19 to 1.05]

14. Secondary Outcome: Change From Baseline to Week 12 in CGI-S Score
Description: as for outcome 3
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for CGI-S score was based on the 83 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 83
units on a scale | 0.00 [-0.14 to 0.14]

15. Secondary Outcome: Change From Baseline to Week 12 in QLS Total Score
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for QLS total score was based on the 82 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | 2.08 [-0.80 to 4.97]

16. Secondary Outcome: Change From Baseline to Week 12 in the 'Common Objects and Activities' QLS Domain Score
Description: as for outcome 5
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for 'Common Objects and Activities' QLS domain score was based on the 82 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | 0.10 (1.16)

17. Secondary Outcome: Change From Baseline to Week 12 in the 'Intrapsychic Foundations' QLS Domain Score
Description: as for outcome 6
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for 'Intrapsychic Foundations' QLS domain score was based on the 82 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | 0.73 (4.31)

18. Secondary Outcome: Change From Baseline to Week 12 in the 'Interpersonal Relations' QLS Domain Score
Description: as for outcome 7
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for 'Interpersonal Relations' QLS domain score was based on the 82 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | 0.67 (4.83)

19. Secondary Outcome: Change From Baseline to Week 12 in the 'Instrumental Role' QLS Domain Score
Description: as for outcome 8
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for 'Instrumental Role' QLS domain score was based on the 81 patients who had a measure for this outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 81
units on a scale | 0.02 (2.53)

20. Secondary Outcome: Change From Baseline to Week 12 in the TooL Total Score
Description: as for outcome 9
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for TooL total score was based on the 82 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | -0.16 [-0.85 to 0.53]

21. Secondary Outcome: Change From Baseline to Week 12 in the WoRQ Total Score
Description: as for outcome 10
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for WoRQ total score was based on the 82 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | -0.55 [-1.20 to 0.11]

22. Secondary Outcome: Change From Baseline to Week 12 in ASEX Total Score
Description: as for outcome 11
Time Frame: Baseline and Week 12
Population: Effectiveness data is based on all patients who received at least one dose of IMP in Study 14724B (APTS). Effectiveness was measured at Weeks 0, 12, and 24. At Week 12, the analysis for ASEX total score was based on the 82 patients who had a measure for this outcome
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
units on a scale | -0.74 [-2.03 to 0.56]

23. Secondary Outcome: Patients Categorised As Sexually Dysfunctional Measured at Week 12 on the ASEX Scale
Description: as for outcome 12
Time Frame: Week 12
Population: This analysis is based on all patients who received at least one dose of IMP in Study 14724B (APTS). At Week 12, the analysis for the number of patients categorised as sexually dysfunctional was based on the 82 patients who had a measure for this outcome
Measure: Number; unit: participants
Arm/Group | Aripiprazole Once-monthly
Number analyzed (Participants) | 82
participants | 32

ADVERSE EVENTS:
Time Frame: Treatment to end of study (up to 28 weeks)
Description: Treatment-Emergent Adverse Events are reported in this section
Arm/Group | Aripiprazole Once-monthly
Serious Adverse Events (participants affected / at risk) | 3/88
Other Adverse Events (participants affected / at risk) | 6/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole Once-monthly (N=88)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Dysphoria (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole Once-monthly (N=88)
Weight increased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No